CLINICAL TRIAL: NCT03765385
Title: The Umeå High-Intensity Training Study: Feasibility and Effect of High-Intensity Training in Older Sedentary People
Brief Title: The Umeå High-Intensity Training Study
Acronym: Umeå HIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dnr 2018-307-31M
Record Dates: First submitted 2018-11-26; First posted 2018-12-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Aged
Keywords: Aged; Aged, 80 and over; Exercise
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome assessors will be masked to group allocation. The participants will be given repeated instructions not to reveal their group allocation to the outcome assessors. Data set will be blinded regarding group allocation (and the code for the groups will be held by a researcher not involved in the study) when performing analyses for main outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity training (Experimental): Each high-intensity training (HIT) session will consist of 10 repeated 6-seconds regulated high intensity cycling sprints against an individualized load set to reach a supramaximal exercise intensity (i.e. power output is higher than power output at maximum oxygen uptake). Session duration for HIT is 20 min, including warm-up and cool-down. The protocol enables controlled and systematic adjustments of training intensity by means of standardized criteria.
  Interventions: Other: High-intensity training
- Moderate-intensity continuous training (Active Comparator): Each moderate-intensity continuous training (MICT) session will consist of aerobic training regulated against an individualized load set to reach a moderate submaximal exercise intensity (i.e. power output is lower than power output at maximum oxygen uptake). Session duration for MICT is 40 min, including warm-up and cool-down. The protocol enables controlled and systematic adjustments of training intensity by means of standardized criteria.
  Interventions: Other: Moderate-intensity continuous training

INTERVENTIONS:
Other: High-intensity training — Sessions will be performed twice weekly for 12 weeks, in groups of 8-10 participants and two supervisors.
  Arms: High-intensity training
Other: Moderate-intensity continuous training — Sessions will be performed twice weekly for 12 weeks, in groups of 8-10 participants and two supervisors.
  Arms: Moderate-intensity continuous training

SUMMARY:
This randomized controlled trial will evaluate the effect of high-intensity training (HIT) in older sedentary people. Seventy older people, aged 65 and over, will be randomized to HIT or moderate-intensity continuous training (MICT). HIT sessions will consist of 10 repeated 6-seconds regulated high intensity cycling sprints against an individualized load. MICT (control group) sessions will consist of aerobic training regulated against an individualized load set to reach a moderate submaximal exercise intensity. Both groups will be performed twice weekly for 12 weeks. The study will evaluate the effects on 1) Cardiovascular function, 2) Brain health, 3) Muscular function, 4) Psychological health, 5) Physical activity, 6) Metabolic health, and 7) Examine the feasibility (attendance, achieved intensity, adverse events) as well as the experiences of HIT. Most outcomes will be assessed at baseline, 3 months (directly after intervention period), and 9 months by blinded assessors.

DETAILED DESCRIPTION:
Information about modifications of the study protocol (September 2020): Experiences of exercising and its effects were at the 9-month follow-up collected through individual interviews instead of focus group interviews (secondary outcome measures no. 31). Due to Covid-19, at the 9-month follow-up all outcome measurements besides the questionnaire (secondary outcome measures no 9, 10, 11, 12, and 14) and interviews (secondary outcome measure no 31) were terminated for 37 of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Not regularly physically active at moderate or high intensity over the last year.
* Independent in activities of daily living (ADL) and able to transfer from home to exercise facility.

Exclusion Criteria:

* Chronic and progressive neurological diseases.
* Movement related conditions and functions (e.g. pain) or heart and lung conditions and diseases that prohibit exercise or tests, based on screening by a physician.
* Cognitive impairment (Mini-Mental State Examination score below 27)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline cardiovascular capacity at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Maximum oxygen uptake (VO2 max)
Change from baseline cognitive function at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Measured using standardized tests covering: episodic memory (free recall, paired associates), executive functions (n-back, Trail Making Test (TMT) 4, flanker task), visuospatial ability (spatial relations), working memory (digit span) and processing speed (Trail Making Test (TMT) 2 and 3). The cognitive tasks are first z-transformed and then everaged to form a unit-weighted cognitive score as well as domain specific constructs.

SECONDARY OUTCOMES:
Change from baseline brain function at 3 months. | Baseline, 3 months
  Assessed using functional MRI (fMRI) using two paradigms. Test A will estimate functional brain response during working memory manipulation and maintenance. Test B will estimate brain response during a pattern completion/separation paradigm. Separate analyses will be performed for fMRI paradigm A and B respectively. For each paradigm changes of % signal BOLD change will be analysed.
Change from baseline brain structure at 3 months. | Baseline, 3 months
  Assessed using standard MRI-sequences including T1w, T2w, T2-FLAIR. For structural MRI data volume (mm3) and cortical thickness (mm) will be the unit of measure.
Change from baseline strength in knee extensors at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Maximal isometric strength in knee extensor measured as normalized joint torque in newton meters per kilogram bodyweight (Nm/kg).
Change from baseline hand grip strength at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Maximal hand grip strength measured as normalized force in Newtons per kilogram bodyweight (N/kg).
Change from baseline leg extensor muscle power at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Leg extensor power in the Nottingham Power Rig, measured as peak power output (watt).
Change from baseline functional performance at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Chair-stand test, number of chair-stands during 30 seconds.
Change from baseline functional balance at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  One-leg stance: number of seconds able to stand on one leg (maximum 120 seconds).
Change from baseline functional balance at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Step test, number of steps during 30 seconds.
Change from baseline anxiety and depression at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Hospital anxiety and depression scale (HAD): range 0-42, higher score indicates more symptoms.
Change from baseline health related quality of life at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Short Form Health Survey (SF-36): scores transformed to 0 to 100, higher scores indicates better quality of life.
Change from baseline self-efficacy at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Swedish Exercise Self Efficacy Scale (ESES-S): Range 10-40, higher score indicates more self efficacy.
Change from baseline sleep quality at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  One question (no. 3) regarding sleep from Montgomery-Åsberg Depression Rating Scale (MADRS).
Change from baseline objective physical activity at 1.5 months (mid-training), at 3 months and at 9 months, respectively. | Baseline, 1.5 months, 3 months, 9 months
  Physical activity measured by an activity monitor, the Actigraph. Number of steps per day and number of activity counts per day will be measured.
Change from baseline self-reported physical activity at 1.5 months (mid-training), at 3 months and at 9 months, respectively. | Baseline, 1.5 months, 3 months, 9 months
  Two indicator questions on physical activity from the Swedish National Board of Health and Welfare.
Change from baseline metabolic health at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Oral glucose tolerance test (OGTT):blood glucose in mmol/l,
Change from baseline lipid profile at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Lipid profile, measured by total cholesterol as well as separately as LDL- cholesterol and HDL-cholesterol. Unit of measure is mmol/l.
Change from baseline inflammation markers at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  C-reactive protein (CRP) in blood sample, units of measure is mg/l.
Change from baseline inflammation markers at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Interleukins in blood sample, units of measure is pg/ml.
Change from baseline neurotrophic factors at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Insulin-like growth factor 1 (IGF-1), units of measure is pg/ml.
Change from baseline neurotrophic factors at 3 months and at 9 months, respectively. | Baseline, 3 months, 9 months
  Brain-derived neurotrophic factor (BDNF), units of measure is pg/ml.
Change from baseline blood pressure at 1.5 months (mid-training), at 3 months and at 9 months, respectively. | Baseline, 1.5 months, 3 months, 9 months
  Blood pressure at rest, measured as systolic ans diastolic pressure in mmHg.
Change from baseline resting heart rate at 1.5 months (mid-training), at 3 months and at 9 months, respectively. | Baseline, 1.5 months, 3 months, 9 months
  Resting heart rate, measured as beats per minute.
Change from baseline autonomic function at 1.5 months (mid-training), at 3 months and at 9 months, respectively. | Baseline, 1.5 months, 3 months, 9 months
  Heart rate variability (HRV), measured in the time domain (e.g. RMSSD) and frequency domain (LF:HF).
Applicability of the interventions | Through the whole 3-month intervention period
  Attendance: number of sessions attended.
Applicability of the interventions | Through the whole 3-month intervention period
  Absolute work-load during training in Watt.
Applicability of the interventions | Through the whole 3-month intervention period
  Relative training intensity, as percentage of MAP (Maximum Aerobic Power output).
Applicability of the interventions | Through the whole 3-month intervention period
  Relative training intensity, as percentage of MHR (maximum heart rate).
Applicability of the interventions | Through the whole 3-month intervention period
  Perceived exertion during training, measured with the Borg Rating of perceived exertion scale (RPE)
Applicability of the interventions | Through the whole 3-month intervention period
  Adverse events, discomfort or chest pain during training measured with the Borg Category ratio scale (CR-10).
Applicability of the interventions | Through the whole 3-month intervention period
  Affective state during training session using Feeling Scale, range -5 to 5, higher score indicates better feeling.
Experiences of exercising and its effects | 3 months, 9 months.
  Focus group interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rosendahl, Professor, Principal Investigator — Umeå University; Carl-Johan Boraxbekk, Professor, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simonsson E, Levik Sandstrom S, Hedlund M, Holmberg H, Johansson B, Lindelof N, Boraxbekk CJ, Rosendahl E. Effects of Controlled Supramaximal High-Intensity Interval Training on Cardiorespiratory Fitness and Global Cognitive Function in Older Adults: The Umea HIT Study-A Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2023 Aug 27;78(9):1581-1590. doi: 10.1093/gerona/glad070. PMID 36972981